CLINICAL TRIAL: NCT00835783
Title: PET/CT in Infection and Inflammation Imaging: Current Utility and Future Perspectives (The PIN-UP Study)
Brief Title: Validation Study of Combined Positron Emission Tomography/Computer Tomography to Diagnose Infection and Inflammation
Acronym: PIN-UP
Status: Terminated | Type: Observational
Why Stopped: Study logistics proved difficult and enrollment never moved beyond the pilot phase.
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Søren Hess, MD, MD, Odense University Hospital
Other Study IDs: 105-K20
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Bacterial Infections; Bacteremia; Gram-Positive Bacterial Infections; Inflammation
MeSH Terms: conditions — Bacterial Infections; Bacteremia; Gram-Positive Bacterial Infections; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- FUO: Patients with fever of unknown origin undergoing FDG-PET/CT as part of work-up.
- BUO: Patients with bacteremia of unknown origin undergoing FDG-PET/CT as part of work-up.
- VGI: Patients with vascular graft infections undergoing FDG-PET/CT as part of work-up.

SUMMARY:
The overall aim is to validate the current use of FDG PET/CT for the diagnosis of infection and inflammation and examine the usefulness of PET/CT applying also other tracers.

The results should allow us to confirm our primary hypothesis: "FDG-PET/CT is better than established methods to confirm or exclude the diagnosis of infection/inflammation".

DETAILED DESCRIPTION:
The study include several part projects, each contributing to the evaluation of the value of FDG-PET/CT in the diagnosis of infection and inflammation. The aims are to establish the diagnostic value in terms of sensitivity, specificity, positive and negative predictive values, interobserver and intraobserver variation.

Part project A FDG-PET/CT in patients with blood culture positive for staphylococcus aureus and unresolved origin of infection.

Part project B FDG-PET/CT in patients with fever of unknown origin.

Part project C FDG-PET/CT in patients suspected of vascular graft infection.

Additionally, we wish to establish an optimal imaging protocol (necessity of fasting, consequences of antibiotic therapy prior to imaging, and the need of contrast), interpretation criteria, and the value of standard uptake values (SUV).

ELIGIBILITY:
Inclusion Criteria:

Part project A

• Blood culture positive for staphylococcus aureus and unresolved origin of infection.

Part project B

* Fever of unknown origin
* Referred for FDG-PET/CT at the Department of Nuclear Medicine, Odense University Hospital.

Part project C

* Suspected vascular graft infection
* Referred for FDG-PET/CT at the Department of Nuclear Medicine, Odense University Hospital.

Exclusion Criteria:

* Patients incapable of giving, refusing or revoking consent
* Patients less than 18 years of age
* Patients from other regions than the Region of Southern Denmark
* Patients who cannot cooperate to PET/CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are referred for FDG-PET/CT at the Department of Nuclear Medicine, Odense University Hospital. Patients are recruited for part project A from the entire hospital through a project nurse at the Department of Infectious Diseases. Patients are recruited for part project B and part project C among all patients referred for FDG-PET/CT as per usual guidelines.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | During diagnostic workup
  Diagnostic parameters of FDG-PET/CT (ie. sensitivity, specificity, positive and negative predictive values, accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Hess, MD, Principal Investigator — Odense University Hospital, Dept. of Nuclear Medicine
Locations (1):
- Odense University Hospital, Dept. of Nuclear Medicine, Odense, Denmark